CLINICAL TRIAL: NCT04136366
Title: The GUARD Trial - Part 1: A Phase 3 Clinical Trial of Repeated Intravitreal Injections of ADX-2191 Versus Standard-of-Care for Prevention of Proliferative Vitreoretinopathy
Brief Title: The GUARD Trial - Part 1: A Phase 3 Clinical Trial for Prevention of Proliferative Vitreoretinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADX-2191-PVR-001
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-10

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: ADX-2191; recurrent retinal detachment; open globe injury
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-2191 (intravitreal methotrexate 0.8%) (Experimental): ADX-2191 (intravitreal methotrexate 0.8%) administered over 16 weeks.
  Interventions: Drug: ADX-2191 (intravitreal methotrexate 0.8%)
- Standard surgical care procedure (Active Comparator): Standard procedure performed.
  Interventions: Other: Standard surgical care procedure

INTERVENTIONS:
Drug: ADX-2191 (intravitreal methotrexate 0.8%) — ADX-2191 (intravitreal methotrexate 0.8%) injected 13 times over 16 weeks upon completion of pars plana vitrectomy
  Arms: ADX-2191 (intravitreal methotrexate 0.8%)
Other: Standard surgical care procedure — Standard surgical care performed upon completion of pars plana vitrectomy
  Arms: Standard surgical care procedure

SUMMARY:
The GUARD Trial is a multi-center, randomized, controlled, adaptive Phase 3 clinical trial of repeated intravitreal injections of ADX-2191 versus standard-of-care for the prevention of proliferative vitreoretinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older of any gender or race
2. Subject is undergoing pars plana vitrectomy due to recurrent retinal detachment due to proliferative vitreoretinopathy or open globe injury
3. Subject is willing and able to provide written informed consent, comply with clinical trial procedures, and return for all clinical trial visits
4. Subjects of childbearing potential must agree to use two forms of birth control for the duration of the clinical trial

Exclusion Criteria:

1. History of severe non-proliferative or proliferative diabetic retinopathy
2. Other planned eye surgery during the course of the trial
3. Participation in a clinical trial with an investigational medicinal product or investigational device within 90 days of subject enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Florida Retina Institute, Orlando, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Emory Eye Center, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Vitreo-Retinal Surgery, Minneapolis, Minnesota
  - Mayo Clinic Ophthalmology, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Long Island VitreoRetinal Consultants, Forest Hills, New York
  - Duke Health Center, Durham, North Carolina
  - OHSU Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Consultants of Houston, Houston, Texas
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- ADX-2191: ADX-2191 (intravitreal methotrexate 0.8%) injected thirteen times over sixteen weeks
- Standard Surgical Care: Standard surgical care performed
Period: Overall Study
Arm/Group | ADX-2191 | Standard Surgical Care
Started | 68 | 38
Completed | 52 | 32
Not Completed | 16 | 6

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- ADX-2191: ADX-2191 (intravitreal methotrexate 0.8%) injected thirteen times over sixteen
- Total: Total of all reporting groups
Arm/Group | ADX-2191 | Standard Surgical Care | Total
Number analyzed (Participants) | 68 | 38 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 23 | 73
  >=65 years | 18 | 15 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 24 | 75
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 60 | 35 | 95
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 58 | 32 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 68 | 38 | 106

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Retinal Detachment Compared to Historical Rates
Description: Percentage of subjects with recurrent retinal detachments requiring reoperation compared to historical rates
Time Frame: Efficacy assessment period (Week 1 to Week 24)
Population: Modified Intent-to-treat population
Measure: Number; unit: percentage of subjects
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 64 | 34
percentage of subjects | 18.8 | 20.6

2. Secondary Outcome: Number of Subjects With Recurrent Retinal Detachment
Description: Number of subjects with recurrent retinal detachment due to proliferative vitreoretinopathy
Time Frame: Efficacy assessment period (Week 1 to Week 24)
Population: Modified Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 64 | 34
Participants | 12 | 7

3. Secondary Outcome: Best-corrected Visual Acuity
Description: Change from baseline of best-corrected visual acuity using an early treatment diabetic retinopathy study (ETDRS) chart. The ETDRS chart contains seventy letters and the visual acuity letter score is equal to the total number of letters read correctly (0 = worst outcome, 70 = best outcome).
Time Frame: Efficacy assessment period (Week 1 to Week 24)
Population: Modified Intent-to-treat population
Measure: Mean (Standard Deviation); unit: correct letters
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 62 | 31
correct letters | 16.9 (23.2) | 22.5 (27.4)

4. Secondary Outcome: Macular Epiretinal Membrane
Description: Number of subjects with macular epiretinal membrane assessed by spectral domain optical coherence tomography for study eye
Time Frame: Week 24
Population: Modified Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 64 | 34
Participants | 18 | 12

5. Secondary Outcome: Intraocular Pressure Less Than 5 mmHg for Study Eye
Description: Number of subjects with intraocular pressure less than 5 mmHg for study eye
Time Frame: Week 24
Population: Modified Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 64 | 34
Participants | 2 | 4

6. Secondary Outcome: Central Macular Subfield Thickness
Description: Number of subjects with central macular subfield thickness assessed by spectral domain optical coherence tomography for study eye
Time Frame: Week 24
Population: Modified Intent-to-treat population
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ADX-2191 | Standard Surgical Care
Number analyzed (Participants) | 64 | 34
microns | 384.4 (185.24) | 473.7 (228.95)

ADVERSE EVENTS:
Time Frame: The safety assessment period was up to twenty-four weeks.
Arm/Group | ADX-2191 | Standard Surgical Care
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/38
Other Adverse Events (participants affected / at risk) | 39/68 | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-2191 (N=68) | Standard Surgical Care (N=38)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-2191 (N=68) | Standard Surgical Care (N=38)
Punctate keratitis (Eye disorders) | 11 (15) | 1 (1)
Eye pain (Eye disorders) | 9 (9) | 9 (10)
Keratitis (Eye disorders) | 6 (12) | 2 (3)
Cystoid macular oedema (Eye disorders) | 5 (5) | 5 (6)
Eye irritation (Eye disorders) | 5 (7) | 0 (0)
Cataract (Eye disorders) | 4 (5) | 3 (4)
Cataract subcapsular (Eye disorders) | 4 (6) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 4 (4) | 3 (3)
Corneal oedema (Eye disorders) | 4 (4) | 4 (4)
Dry eye (Eye disorders) | 4 (4) | 2 (2)
Macular fibrosis (Eye disorders) | 4 (4) | 6 (6)
Vision blurred (Eye disorders) | 4 (4) | 1 (1)
Anterior chamber inflammation (Eye disorders) | 3 (4) | 3 (3)
Macular Oedema (Eye disorders) | 3 (4) | 3 (3)
Corneal epithelium defect (Eye disorders) | 2 (2) | 4 (4)
Anterior chamber cell (Eye disorders) | 1 (1) | 4 (6)
Hypotony of eye (Eye disorders) | 1 (1) | 2 (2)
Iris adhesions (Eye disorders) | 1 (1) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Anterior chamber fibrin (Eye disorders) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2)
Posterior capsule opacification (Eye disorders) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 5 (6) | 2 (3)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Intraocular pressure increased (Investigations) | 2 (2) | 8 (9)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04136366/Prot_SAP_000.pdf